CLINICAL TRIAL: NCT03712553
Title: Behavioral Science and Hepatitis C Screening Outreach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Shivan J Mehta, Assistant Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 831526
Record Dates: First submitted 2018-10-16; First posted 2018-10-19 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Hepatitis C
Keywords: Behavioral Economics; Screening; Outreach
MeSH Terms: conditions — Hepatitis C | interventions — College Fraternities and Sororities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- A1: Opt-In, UC Letter (Active Comparator): Behavioral: Opt-In vs. Opt-Out The usual care (UC) letter consists of an opt-in message encouraging participants to contact their primary care provider for Hepatitis C screening.
  Interventions: Behavioral: Letter; Behavioral: Usual Care Messaging
- A2: Opt-Out, UC Letter (Experimental): Behavioral: Opt-In vs. Opt-Out The usual care (UC) letter consists of a message and a written laboratory order from primary care provider to complete Hepatitis C screening.
  Interventions: Behavioral: Opt-Out; Behavioral: Usual Care Messaging
- B1: Active MPM User, UC Letter (Experimental): Behavioral: Letter vs. Electronic Messaging Behavioral: Usual Care Messaging vs. Behavioral Economic Messaging Participants who are active MyPennMedicine (MPM) users receive a usual care (UC) letter consisting of a message encouraging them to contact their primary care provider for Hepatitis C screening.
  Interventions: Behavioral: Letter
- B2: Active MPM User, BE Letter (Experimental): Behavioral: Letter vs. Electronic Messaging Behavioral: Usual Care Messaging vs. Behavioral Economic Messaging Participants who are active MyPennMedicine (MPM) users receive a letter with behavioral economic (BE) principles encouraging them to contact their primary care provider for Hepatitis C screening.
  Interventions: Behavioral: Letter; Behavioral: Behavioral Economic Messaging
- B3: Active MPM User, UC MPM Message (Active Comparator): Behavioral: Letter vs. Electronic Messaging Behavioral: Usual Care Messaging vs. Behavioral Economic Messaging Participants who are active MyPennMedicine (MPM) users receive an electronic usual care (UC) message on the MyPennMedicine patient portal encouraging them to contact their primary care provider for Hepatitis C screening.
  Interventions: Behavioral: Usual Care Messaging
- B4: Active MPM User, BE MPM Message (Experimental): Behavioral: Letter vs. Electronic Messaging Behavioral: Usual Care Messaging vs. Behavioral Economic Messaging Participants who are active MyPennMedicine (MPM) users receive an electronic message with behavioral economic principles on the MyPennMedicine patient portal encouraging them to contact their primary care provider for Hepatitis C screening.
  Interventions: Behavioral: Behavioral Economic Messaging
- B5: Non-MPM User, UC Letter (Active Comparator): Behavioral: Usual Care Messaging vs. Behavioral Economic Messaging Participants who are non-MyPennMedicine (non-MPM) users receive a usual care (UC) letter consisting of a message encouraging them to contact their primary care provider for Hepatitis C screening.
  Interventions: Behavioral: Letter; Behavioral: Usual Care Messaging
- B6: Non-MPM User, BE Letter (Experimental): Behavioral: Usual Care Messaging vs. Behavioral Economic Messaging Participants who are non-MyPennMedicine (non-MPM) users receive a letter with behavioral economic principles (BE) encouraging them to contact their primary care provider for Hepatitis C screening.
  Interventions: Behavioral: Letter; Behavioral: Behavioral Economic Messaging

INTERVENTIONS:
Behavioral: Opt-Out — Opt-In messaging prompts participants to contact their primary care provider to receive Hepatitis C screening whereas Opt-Out messaging includes a signed laboratory order for Hepatitis C screening.
  Arms: A2: Opt-Out, UC Letter
Behavioral: Letter — Participants receive messaging prompting them to contact their primary care provider to receive Hepatitis C screening, either as a letter or an electronic message on the MyPennMedicine patient portal.
  Arms: A1: Opt-In, UC Letter; B1: Active MPM User, UC Letter; B2: Active MPM User, BE Letter; B5: Non-MPM User, UC Letter; B6: Non-MPM User, BE Letter
Behavioral: Behavioral Economic Messaging — Participants receive standard messaging about HCV and ways to get screened and messaging that incorporates behavioral economic principles such as norms, reciprocity, anticipated regret, and pre-commitment to get screening.
  Arms: B2: Active MPM User, BE Letter; B4: Active MPM User, BE MPM Message; B6: Non-MPM User, BE Letter
Behavioral: Usual Care Messaging — Participants receive standard messaging about HCV and ways to get screening.
  Arms: A1: Opt-In, UC Letter; A2: Opt-Out, UC Letter; B3: Active MPM User, UC MPM Message; B5: Non-MPM User, UC Letter

SUMMARY:
This project aims to evaluate different approaches to increase Hepatitis C screening among primary care patients at Penn Medicine through a centralized screening outreach program. In a pragmatic trial, we will evaluate different approaches to increase completion of screening among eligible patients, including changing the default from opt-in to opt-out and incorporating behavioral science principles into the outreach communication.

DETAILED DESCRIPTION:
The hepatitis C virus (HCV) is the leading cause of liver transplant and hepatocellular carcinoma in the US. New direct-acting antivirals are available that can eradicate the disease in over 95% of those that are treated, with minimal side effects. As a result of new therapies and a five-fold higher risk among baby boomers, the US Preventive Services Task Force and CDC now recommend HCV screening for all patients born between 1945 and 1965. Of the estimated 3.2 million people chronically infected with HCV, about 75% were born during this time frame. Despite this, national rates of screening among this group remain low at less than 30%. If more people could get screened, we could potentially identify more undiagnosed disease and help navigate to treatment.

At Penn Medicine primary care practices, HCV screening rates have risen from 37% in 2014 to 61% in 2017, likely from a combination of provider educational efforts and EHR alerts. There is also significant practice variation ranging from 4% to 99% screening rates. While EHR alerts have been shown to increase HCV screening rates, there is potential to complement this with direct outreach to patients homes, as has been incorporated into cancer screening initiatives. Additionally, there is a mandate from the state of Pennsylvania requiring health care providers to offer HCV testing to all primary care patients. There is an opportunity to provide direct outreach to all eligible primary care patients at Penn Medicine, while also evaluating different approaches to increasing HCV screening rates.

Insights from behavioral science have been shown to increase participation in health promoting behaviors in a variety of ways. Switching from opt-in to opt-out framing has been shown to triple patient participation in remote monitoring and CRC screening. Additionally, messaging that incorporates social norms, reciprocity, and precommitment have also been shown to increase participation. However, it is not clear how these approaches would translate to HCV screening.

ELIGIBILITY:
Inclusion Criteria:

* at least 2 visits to primary care provider within 2 years
* born between 1945 and 1965

Exclusion Criteria:

* have had 1 HCV antibody test, viral load test or are considered up-to-date on HCV screening by health maintenance

Ages: 53 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21493 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
HCV Antibody Completion within 4 Months | 4 months
  Percentage of patients who complete HCV antibody testing within 4 months of initial outreach

SECONDARY OUTCOMES:
HCV Antibody Completion within 12 Months | 12 months
  Percentage of patients who complete HCV antibody testing within 12 months of initial outreach
HCV Antibody Positive | 12 months
  Percentage of tests that are positive
HCV Antibody Positive with Viral Loads | 12 months
  Percentage of test that are positive with detectable viral loads
Referred to Specialist | 12 months
  Percentage of patients referred to specialist and receive HCV treatment and cure

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, MBA, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta SJ, Day SC, Norris AH, Sung J, Reitz C, Wollack C, Snider CK, Shaw PA, Asch DA. Behavioral interventions to improve population health outreach for hepatitis C screening: randomized clinical trial. BMJ. 2021 May 18;373:n1022. doi: 10.1136/bmj.n1022. PMID 34006604